CLINICAL TRIAL: NCT06599580
Title: Mother Screening for Relapse Using Mid-upper Arm Circumference Among Children Recovered From Severe Acute Malnutrition (MAMAN)
Brief Title: Mother Screening for Relapse Using Mid-upper Arm Circumference Among Children Recovered From Severe Acute Malnutrition (Full Scale Trial)
Acronym: MAMAN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Centre de Recherche en Sante de Nouna, Burkina Faso (Other Government); Thrasher Research Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 24-42418
Record Dates: First submitted 2024-09-13; First posted 2024-09-19 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Malnutrition, Child; Malnutrition, Infant; Malnutrition or Risk of Malnutrition; Hemoglobin Level Measurement; Anemia
Keywords: MUAC (mid-upper arm circumference); Caregiver screening; malnutrition; home based malnutrition screening
MeSH Terms: conditions — Child Nutrition Disorders; Infant Nutrition Disorders; Malnutrition; Anemia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard of care treatment and follow-up schedule without alteration (control arm) (No Intervention): This arm with serve as the control arm and receive the current standard of care, which is no caregiver training to conduct mid-upper arm circumference screenings and monthly clinic-based follow-up appointments for 3 months with a final visit at 6 months post enrollment.
- Caregiver mid-upper arm circumference (MUAC) screening and a standard of care follow-up schedule (Experimental): This arm will include caregiver screening with a mid-upper arm circumference tape at home weekly. Caregivers will be trained to screen their child for malnutrition relapse using mid-upper arm circumference tapes and requested to bring their child back to the clinic when relapse is detected. Additionally, this arm will receive the standard of care, which includes a monthly follow-up schedule for the first 3 months post enrollment and a final follow-up at 6 months.
  Interventions: Behavioral: Training caregivers to screen children for malnutrition relapse
- Caregiver mid-upper arm circumference (MUAC) screening and a reduced follow-up schedule (Experimental): This arm will include caregiver screening with a mid-upper arm circumference tape at home weekly. Caregivers will be trained to screen their child for malnutrition relapse using mid-upper arm circumference tapes and requested to bring their child back to the clinic when relapse is detected. Additionally, this arm will receive a reduced follow-up schedule at the clinic, which will include one planned visit at 3 months post enrollment and a final follow-up visit at 6 months.
  Interventions: Behavioral: Training caregivers to screen children for malnutrition relapse; Other: Reduced follow-up schedule

INTERVENTIONS:
Behavioral: Training caregivers to screen children for malnutrition relapse — Caregivers enrolled in the trial who are assigned to the two experimental arms, will be provided mid-upper arm circumference tapes and trained on how to screen their child for malnutrition relapse and asked to bring their child back to the clinic if relapse is detected.
  Other Names: Caregiver and/or mother mid-upper arm circumference screening
  Arms: Caregiver mid-upper arm circumference (MUAC) screening and a reduced follow-up schedule; Caregiver mid-upper arm circumference (MUAC) screening and a standard of care follow-up schedule
Other: Reduced follow-up schedule — Caregivers in one of the caregiver mid-upper arm circumference screening arms, will be asked to adhere to a reduced follow-up clinic visit schedule for when they bring their child to the clinic for planned visits. The standard of care includes monthly visits for the first 3 months post recovery, but those randomized to the reduced follow-up schedule arm, will not bring their child to the clinic for planned visits 1 month and 2 months after baseline.
  Other Names: Reduced clinic visits
  Arms: Caregiver mid-upper arm circumference (MUAC) screening and a reduced follow-up schedule

SUMMARY:
A 1:1:1 individually randomized unmasked controlled trial is proposed in which caregivers will be trained to screen their children who have recovered from an episode of SAM (severe acute malnutrition) using MUAC (mid-upper arm circumference) tapes. One arm will include caregiver screening with a mid-upper arm circumference tape and usual monthly follow-up schedule for the first 3 months post enrollment and a final follow-up at 6 months. Another arm will include caregiver screening with a mid-upper arm circumference tape and a reduced follow-up schedule for one visit at 3 months and a final visit at 6 months. The third arm will adhere to the current standard of care, which is no caregiver training to conduct mid-upper arm circumference screenings and monthly clinic-based follow-up appointments for 3 months with a final visit at 6 months post enrollment. Children aged 6-54 months with a documented recovery from uncomplicated severe acute malnutrition that was managed in a participating outpatient nutritional program and their caregivers will be eligible for inclusion in the trial. Caregivers will be trained to screen their children weekly for 6 months following discharge from the nutritional program and will be counseled to bring their child back to the nutritional program should their mid-upper arm circumference value fall in the red zone of the mid-upper arm circumference tape (< 11.5 cm). All children will be seen at 3 and 6 months for the primary outcome assessment. By conducting this study, our primary goal is to determine if training caregivers to screen their children for relapse to MAM (moderate acute malnutrition) or SAM (severe acute malnutrition) using mid-upper arm circumference tapes following recovery from SAM (severe acute malnutrition) will reduce the risk of relapse. An additional aim is to assess the level of acceptability of caregivers screening children for malnutrition using mid-upper arm circumference tapes from both a clinic and caregiver perspective.

DETAILED DESCRIPTION:
A pilot randomized controlled trial for MAMAN was conducted to find if training caregivers to perform mid-upper arm circumference measurements to screen for malnutrition is feasible. This research will be expanded by assessing caregiver screening for detection of moderate acute malnutrition or severe acute malnutrition relapse with a 1:1:1 randomized controlled trial enrolling caregiver-child dyads of an increased sample size of 1200 dyads, totaling 2400 individuals. This study will address the need for evidence of the effectiveness of caregiver administered mid-upper arm circumference screening in the improvement of outcomes for children who have recovered from severe acute malnutrition. The effectiveness of training caregivers to screen for child malnutrition relapse using mid-upper arm circumference tapes, risk of relapse, speed of relapse detection, and anthropometric outcomes of the children will be analyzed. This will assist in providing evidence to incorporate the routine inclusion of mid-upper arm circumference screening training for all caregivers of children who are being discharged from severe acute malnutrition treatment.

SPECIFIC AIM 1: Determine the effectiveness of training caregivers to screen for relapse to moderate acute malnutrition or severe acute malnutrition using mid-upper arm circumference tapes following recovery from severe acute malnutrition for improving anthropometric outcomes and improving time to relapse detection. It is hypothesized that caregiver screening will be effective for reducing time to detection of relapse and that children receiving caregiver screening will have better anthropometric measures at 6 months post recovery and faster time to detection of relapse among those who relapse.

* Specific Aim 1A: Determine if detection of relapse in children who have recently recovered from severe acute malnutrition is more expeditious when caregivers are trained to screen for relapse to moderate acute malnutrition or severe acute malnutrition using mid-upper arm circumference tapes compared to current standard of care. It is hypothesized that a reduction in time to relapse detection will occur when caregivers are trained to screen for relapse to moderate acute malnutrition or severe acute malnutrition using mid-upper arm circumference tapes.
* Specific Aim 1B: Determine the effectiveness of caregivers screening mid-upper arm circumference measurements on improving anthropometric outcomes for children. It is hypothesized that training for caregiver screening of mid-upper arm circumference will lead to earlier intervention and improved anthropometric outcomes for children at 12 months post-admission.

SPECIFIC AIM 2: Determine the acceptability caregiver mid-upper arm circumference training. It is hypothesized that most survey responses at the 3 and 6-month visits will show high levels of acceptance towards caregiver screening of children using mid-upper arm circumference tapes.

ELIGIBILITY:
Inclusion Criteria:

* Caregiver's aged 18 years old or older or a legal guardian or a relative aged 18 or older
* Child aged 6-54 months
* Child has recovered from an episode of severe acute malnutrition per Burkinabè national guidelines (weight-for-height ≥ -2 and/or mid-upper arm circumference ≥ 12.5 cm in the past month, with the criterion used for admissions corresponding to the original admission criteria)
* Family is planning to stay in the study area for 6 months
* Appropriate consent from the caregiver or guardian.

Exclusion Criteria:

* Caregiver age under 18 years old, or legal guardian or relatives under 18 years old
* Child age < 6 months or > 54 months
* Twins/multiple births
* Children with feeding issues
* Did not recover from severe acute malnutrition in the past month
* Family is planning to move out of the study area in the next 6 months
* Caregiver or guardian refuses to provide consent

Ages: 6 Months to 54 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2400 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of relapse | 6 months
  The primary outcome will be defined as the proportion of children who relapse to global acute malnutrition (either moderate acute malnutrition with mid-upper arm circumference < 12.5 cm to ≥ 11.5 cm and/or weight-for-height Z score < -2 to ≥ -3 or severe acute malnutrition with mid-upper arm circumference < 11.5 cm and/or weight-for-height Z score < -3) by the 6 month primary endpoint randomized by study assignment.

SECONDARY OUTCOMES:
Time to detection of relapse | 6 months
  The amount of time until the detection of malnutrition relapse will be assessed as a secondary outcome and will be defined as the time from the baseline visit until the planned or unplanned visit when malnutrition relapse is detected. This will be measured up until the 6 month visit and will be assessed by randomized study assignment.
Cumulative incidence of relapse to MAM or SAM separately | 6 months
  The proportion of children by randomized allocation who relapse to MAM or to SAM analyzed separately.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Oldenburg, ScD, Principal Investigator — University of California, San Francisco
Locations (1):
- Centre de recherche en sante de nouna, Nouna, Burkina Faso

IPD SHARING:
Plan to Share IPD: No